CLINICAL TRIAL: NCT06029907
Title: Project HOPES: Healthy Options for Pain and Ending Smoking. A Program for Cancer Survivors.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00113492
Record Dates: First submitted 2023-08-23; First posted 2023-09-08 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Smoking Cessation; Pain
Keywords: Smoking cessation; Pain management; Cancer survivors
MeSH Terms: conditions — Smoking Cessation; Pain; Agnosia | interventions — Varenicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Study population (Other): All patients will receive a smoking cessation and pain management intervention combined with clinician-prescribed varenicline.
  Interventions: Other: Smoking cessation and pain management intervention; Drug: Varenicline

INTERVENTIONS:
Other: Smoking cessation and pain management intervention — Patients will receive a behavioral smoking cessation and pain management intervention
Drug: Varenicline — Patients will receive varenicline prescribed by their oncologist
  Other Names: Chantix; Chantix Starting Month Box; Tyrvaya

SUMMARY:
The proposed pilot study will develop and test feasibility, acceptability, and signal for efficacy of a smoking cessation and pain management intervention for 20 cancer survivors.

DETAILED DESCRIPTION:
The proposed pilot study will develop and test feasibility, acceptability, and signal for efficacy of a smoking cessation and pain management intervention for 20 cancer survivors. There are two specific aims:

Aim 1: To test the feasibility and acceptability of a behavioral smoking cessation and pain management intervention combined with varenicline.

Aim 2: To examine the smoking cessation rate and changes in pain (i.e., severity, interference), self-efficacy (i.e., smoking cessation, pain management), and quality of life from baseline to post-intervention and 3-months post-baseline.

The proposed intervention could have a great impact on the health and quality of life of cancer survivors. Teaching pain management techniques coupled with smoking cessation techniques addresses two critical issues for survivors.

The study team submitted an R01 based on a prior pilot study. Reviewers were enthusiastic about the significance and innovation of addressing smoking and pain simultaneously. They were, however, not convinced by the potential efficacy of our pilot data. They suggested the study team test the same intervention with varenicline as it can both help promote smoking cessation and provide some analgesia for pain. To address reviewer concerns to lead to R01 funding, the study team proposes to build on our combined behavioral smoking cessation and behavioral pain intervention by adding varenicline.

BACKGROUND AND SIGNIFICANCE:

The US currently has an estimated 15.5 million cancer survivors. Approximately 10-30% of all cancer survivors are current smokers at diagnosis. Well more than half (70%) of survivors who are current smokers at diagnosis will either resume smoking after an initial quit attempt or continue smoking following their diagnosis. Those who live in rural areas have an even higher rate of smoking. As many as 70% also suffer from pain as well as other physical and/or psychosocial problems. Although some survivors hold beliefs that smoking reduces pain and alleviates distress, in fact, persistent smoking following cancer diagnosis is associated with worse pain, poor quality of life, increased risk for disease recurrence, and worsening of many comorbid medical conditions. Of importance, quitting smoking significantly improves survivors' response to cancer treatment, reduces cancer recurrence, mitigates risk of new cancers and cardiovascular disease and improves quality of life. Thus, helping survivors quit smoking and learn how to manage their pain is a top priority for oncology providers.

To date, integration of best practices for promoting smoking cessation and pain management among cancer survivors has received little attention, despite smokers who experience pain reporting lower self-efficacy for quitting and greater expectancies of severe withdrawal and poor cessation outcomes. Building upon our longstanding expertise in smoking cessation and pain management interventions, the study team proposes to build on our pilot work by including a pharmacologic agent that can enhance both cessation and pain management. Among pharmacologic treatments, varenicline (i.e., Chantix) has the strongest evidence for helping people quit smoking. Varenicline also acts on receptors to potentially block pain. The study team submitted an R01, and reviewers wanted stronger pilot data that convinced them more that combining a smoking cessation and pain management intervention would help survivors quit smoking. Thus, in addition to published pilot data the study team have with cancer survivors recruited from the Duke Cancer Network (DCN), the study team proposes to recruit survivors who smoke to test whether the study team can increase our cessation rate by adding varenicline to our behavioral smoking cessation pain management program. In our prior pilot, the study team found promising evidence for the feasibility, acceptability, and signal for efficacy of a combined behavioral smoking cessation with nicotine replacement patches and behavioral pain management intervention. Survivors who received the intervention rated it as useful for smoking cessation and pain management. Survivors who received the intervention were more likely to quit smoking than those in the control arm, but only a few survivors quit. Survivors in the intervention compared to the control arm reported improvements in their pain as well as depression and physical well-being, but again these changes were small. Thus, in this proposed pilot, the study team will examine whether adding varenicline to our behavioral program helps more survivors quit smoking and report better pain management. Our primary outcomes will be feasibility, acceptability, and evidence for potential of future efficacy testing a new combination of behavioral smoking cessation and behavioral pain management + varenicline. Our secondary outcome will be biochemically verified 7-day point prevalence smoking abstinence at 3 months. The study team will also examine pain, self-efficacy (smoking, pain management), and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer at our targeted recruitment sites
* Have a diagnosis of cancer within the past 5 years (can be currently undergoing treatment)
* Have a life expectancy of at least 1 year
* Report pain within the last 3 weeks of 3 or higher on a 10 point scale
* Have smoked at least 100 cigarettes in their lifetime
* Smoke 5 or more cigarettes per day in the prior 7 days
* Be willing to try to quit smoking
* Not participating in another smoking cessation trial
* Age 18 or older
* Speak English

Exclusion Criteria:

* Hearing impaired
* Deemed too sick to participate
* Evidence of unstable cognitive or mental health problems who cannot properly provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Number of patients who complete the study | through study completion, an average of 1 year
  Completing study participation is the number of those who attend all sessions and complete follow-up surveys. This will serve as our feasibility benchmark.
Number of patients who report that the intervention was helpful | through study completion, an average of 1 year
  Patients will be asked if they found the intervention helpful on follow-up surveys. This will serve as our acceptability benchmark.

SECONDARY OUTCOMES:
Number of Patients at 3-month Post-Intervention with Validated Cessation | through study completion, an average of 1 year
  Biochemically verified 7-day point prevalence smoking abstinence at 3 months with use of CO monitors.
Change in patient-reported pain (severity, interference) | through study completion, an average of 1 year
  Patients will report their pain on a scale from 0-10 [0 being "no pain" and 10 being "pain as bad as you can imagine"] and report how pain is affecting their lives 0-10 [0 being "does not interfere" and 10 being "completely interferes"] on administered surveys at baseline, post-intervention, and 3-month post-intervention. Study team will look to see if there is a change in patient-reported pain.
Change in patient-reported self efficacy (smoking cessation, pain management) | through study completion, an average of 1 year
  Patients will report their ability to stop smoking and manage their pain on administered surveys at baseline, post-intervention, and 3 month-post intervention. Self-efficacy is measured on a scale from 1 to 7 where 1 is "not confident at all" and 7 is "extremely confident". Pain management is measured on a scale of 1-10 where 1 is "very uncertain, 5 is "moderately uncertain", and 10 is "very uncertain". Study team will look to see if there is a change in patient-reported self efficacy
Change in patient-reported quality of life (Depression/Mood/Negative Affect) | through study completion, an average of 1 year
  Patients will respond to questions about their perceived quality of life on administered surveys at baseline, post-intervention, and 3 month post-intervention. Quality of life will be measured based on questions related to Depression/Mood/Negative Affect (Hospital Anxiety Depression Scale - HADS). The HADS is comprised of two sub scales, Depression and Anxiety. Each subscale has a score ranging from 0-21.Items are rated on a 4-point Likert-type scale ranging from 0 t o 3, generating a scale range of 0 to 42 points, with higher scores representing greater symptom severity. The anxiety subscale has 3 items that refer to panic and 4 to generalized anxiety. Add the A questions to get a score for anxiety and the D questions for depression. Scores of 0-7 indicate normal levels of anxiety and depression; 8-10 indicate borderline abnormal anxiety. Study team will look to see if there is a change in patient-reported quality of life.
Change in patient-reported quality of life (Coping) | through study completion, an average of 1 year
  Patients will respond to questions about their perceived quality of life on administered surveys at baseline, post-intervention, and 3 month post-intervention. Quality of life will be measured based on questions related to Coping. Patients will answer questions on scale from "never", "seldom", "occasionally", "often", or "most of the time". Subscale of the Rhode Island Stress and Coping Inventory. Study team will look to see if there is a change in patient-reported quality of life.
Change in patient-reported quality of life (Physical Well Being) | through study completion, an average of 1 year
  Patients will respond to questions about their perceived quality of life on administered surveys at baseline, post-intervention, and 3 month post-intervention. Quality of life will be measured based on questions related to Physical Well Being. Patients will answer questions on a 5-point scale from "0: not at all", "1: a little bit", "2: somewhat", "3: quite a bit", or "4: very much". Study team will look to see if there is a change in patient-reported quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn I Pollak, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No